CLINICAL TRIAL: NCT07286942
Title: Stereotactic Body Radiotherapy With Sequential Iparomlimab and Tuvonralimab (QL1706) + Chemotherapy as Neoadjuvant Therapy in Patients With Resectable Non-small-cell Lung Cancer in China (LUNG-Nanjing01): a Single-arm, Single-centre, Phase 2 Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Zhang Zhi, Associate Professor, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUNG-Nanjing 01
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: NSCLC; NSCLC (Non-small Cell Lung Cancer)
Keywords: NSCLC; SBRT; neoadjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant SBRT in combination with apalolimab and toripalimab (QL1706) plus (Experimental)
  Interventions: Drug: apalolimab and toripalimab (QL1706)

INTERVENTIONS:
Drug: apalolimab and toripalimab (QL1706) — QL1706 is a bispecific antibody developed using the MabPair™ biotechnology platform. It comprises two engineered monoclonal antibodies targeting PD-1 and CTLA-4, respectively, in a fixed ratio of approximately 2:1 (65:35 ± 10%).

SUMMARY:
The primary objective of this study is to evaluate whether neoadjuvant SBRT as an immunomodulator in combination with apalolimab and toripalimab (QL1706) plus chemotherapy improves the pathological complete response (pCR) rate in patients with resectable stage IIA-IIIB LUAD. The secondary objectives include major pathological response (MPR), disease-free survival (DFS), R0 resection rate, the feasibility and safety. Moreover, the potential predictors for pathological response also will be explored.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, phase II trial (LUNG-Nanjing01 study), patients will be recruited from Affiliated Cancer Hospital of Nanjing Medical University, Jiangsu, China. Eligible participants are adults aged 18 or older, a biopsy-confirmed diagnosis of locally advanced NSCLC, clinical stage IIA to IIIB (according to the 9th edition of the American Joint Committee on Cancer staging system), determined by computed tomography and/or magnetic resonance imaging before treatments and deemed surgical resectable with curative intent. Every patient will be evaluated by a multidisciplinary team consisting of thoracic surgeons, medical oncologists, radiation oncologists, radiologists, and pathologists. Enrolled patients have no prior cancer treatments, with an Eastern Cooperative Oncology Group performance status of 0 or 1, regardless of smoking history and PD-L1/PD-1 expression.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participates in the study and provides written informed consent;
2. Aged 18-75 years, with no restriction on sex;
3. Histologically or cytologically confirmed diagnosis of non-small-cell lung cancer (NSCLC);
4. Has not received prior systemic therapy and is willing to undergo neoadjuvant treatment for stage cⅡ-Ⅲ (N2a) disease, according to the 9th edition of the AJCC staging system (Appendix 1);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (see Appendix 2 for scoring criteria);
6. Considered by the thoracic surgeon to have adequate pulmonary reserve to tolerate the planned lung resection;
7. Availability of tumor tissue prior to enrollment for pathological confirmation of EGFR/ALK wild-type status and PD-L1 expression assessment;
8. No significant hematologic, cardiac, pulmonary, hepatic, renal, or immunologic dysfunction, with the following laboratory parameters meeting the specified criteria:

   * Bone marrow function: absolute neutrophil count (ANC) ≥1.5×10⁹/L; platelet count ≥80×10⁹/L; hemoglobin ≥9 g/dL;
   * Liver function: total bilirubin ≤1.5× upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5× ULN;
   * Renal function: serum creatinine ≤1.5× ULN or creatinine clearance ≥60 mL/min; blood urea nitrogen ≤200 mg/L;
9. Women of childbearing potential must have a negative serum pregnancy test within 3 days before the first dose of study treatment.

Exclusion Criteria:

* 1. Presence of locally advanced unresectable or metastatic disease. Unresectable disease is defined according to the 2019 Multidisciplinary Consensus on Stage III Non-Small-Cell Lung Cancer (NSCLC), including certain stage IIIA and IIIB cases and all stage IIIC cases. Typically, this includes N2 disease with a single mediastinal lymph node ≥3 cm in short axis or multiple fused lymph nodes (≥2 cm in short axis on CT), as well as T4 lesions invading the esophagus, heart, aorta, or pulmonary veins, and all N3 disease.

  2. Superior sulcus (Pancoast) NSCLC, large-cell neuroendocrine carcinoma (LCNEC), or sarcomatoid carcinoma.

  3. Known EGFR-sensitive mutations or ALK rearrangements (non-squamous participants must have confirmed EGFR and ALK mutation status).

  4. Prior systemic anticancer therapy for early-stage NSCLC, including investigational agents.

  5. Active infection, or unexplained fever >38.5 °C within 2 weeks prior to screening (participants with tumor-related fever, as judged by the investigator, may be enrolled).

  6. Male or female participants of reproductive potential who are unwilling to use effective contraception during the study; pregnant or breastfeeding women.

  7. Any condition that, in the opinion of the investigator, could interfere with study participation or completion, including severe comorbidities (including psychiatric disorders) requiring concurrent treatment, or family or social factors that may compromise participant safety or data integrity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2027-12-18 (Estimated); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
pCR | up to surgery

SECONDARY OUTCOMES:
MPR | up to surgery
DFS | assessments were performed every 3 months during the first 3 years after surgery and every 6 months during years 3-5 of follow-up
Safety(AEs) | All participants were followed for safety until 90 days after the last dose of study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China